CLINICAL TRIAL: NCT06378450
Title: Examining Dose-Response Effects of Mindfulness Meditation Interventions on Wellbeing: A Randomized Controlled Trial
Brief Title: Dose-Response Effects of Mindfulness Meditation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Responsible Party: Principal Investigator, Nicholas Van Dam, Associate Professor, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2022-23892-31512-2
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Well-Being, Psychological; Depression
MeSH Terms: conditions — Psychological Well-Being; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 10-minute dose (Experimental): Daily guided mindfulness meditation practices of 10-minute duration.
  Interventions: Behavioral: Mindfulness meditation guided practice
- 20-minute dose (Experimental): Daily guided mindfulness meditation practices of 20-minute duration.
  Interventions: Behavioral: Mindfulness meditation guided practice
- 30-minute dose (Experimental): Daily guided mindfulness meditation practices of 30-minute duration.
  Interventions: Behavioral: Mindfulness meditation guided practice
- 3-4 minute minimal dose (Active Comparator): Short daily meditation approximating 3-4 minute duration (akin to the breathing space practice in Mindfulness-based Cognitive Therapy or short practices in popular meditation apps).
  Interventions: Behavioral: Mindfulness meditation guided practice

INTERVENTIONS:
Behavioral: Mindfulness meditation guided practice — Participants will listen to recordings of mindfulness meditation practices from a newly developed 28-day program.

SUMMARY:
The goal of this randomized controlled trial is to test for evidence of dose-response effects in a sample of healthy adults with little to no prior experience with meditation.

The main question it aims to answer is whether larger doses of mindfulness meditation yield greater positive changes in wellbeing than smaller doses.

Our hypotheses are that (1) larger doses of mindfulness training will yield significantly larger effects, and (2) different doses will be significantly associated with variation in participant engagement, with lower engagement associated with higher doses.

Researchers will compare each of three dose conditions, 10-min, 20-min, 30-min, against a minimal dose condition of 3-4 min.

Participants will take a 28-day mindfulness meditation course, with guided audio instructions provided daily throughout the intervention period (excluding one rest day per week). They will also be asked to respond to surveys before, during, and after the intervention.

DETAILED DESCRIPTION:
The study will compare the efficacy of receiving different "doses" of mindfulness training over a 28-day period in a prospective 4-armed, parallel-group randomised controlled trial. Participants will be randomised into one of the 4 groups: 10 minutes of meditation per day, 20 minutes of meditation per day, 30 minutes of meditation per day, or a minimal dose of 3-4 minutes of meditation per day. All participants will be encouraged not to complete any further mindfulness training or practice during the intervention period, apart from informal practice during daily life.

Self-reported biopsychosocial measures will be evaluated at four time points; before randomization (baseline; T0), 2 weeks after randomisation (mid-intervention, T0.5), 4 weeks after randomization (post-intervention; T1), and 2 months after randomization (post follow-up; T2). In addition, weekly and daily outcomes will be evaluated between T0 and T1. Individual adherence and meditation-related experiences (including adverse events) will be monitored and compared across treatments. The trial will consist of three main phases: the Run-in Period, the Intervention Period, and the Follow-up period, as described below.

ELIGIBILITY:
Inclusion Criteria:

* Reside in Australia, with no plans to relocate or travel overseas during the intervention period;
* Sufficient comprehension of the English language to complete measures;
* Register for an account and agree to the Terms and Conditions of Unforgettable.Me;
* If suffering anxious or depressive symptoms of moderate severity (defined by > 19 on the Patient-Reported Outcomes Measurement Information System [PROMIS] Level 2 Anxiety or > 22 on the PROMIS Level 2 Depression), must agree to continue recommended routine medical treatment for eligible underlying mental and/or physical health conditions or the duration of the study and to seek additional treatment if indicated by deterioration of symptoms;
* No or minimal experience with meditation, defined as less than 25 hours over the past 6 months; never attended a multi-day mindfulness course (e.g., Mindfulness-Based Stress Reduction, Vipassana). If 50% of our target sample size has not bee recruited within the first three months of active recruitment, the inclusion criteria will be broadened to include participants with up to 100 hours in the past 6 months.

Exclusion Criteria:

* Self-reported current or lifetime serious mental illness (e.g., neurodevelopmental, schizophrenia spectrum, bipolar, obsessive-compulsive, trauma-related, dissociative or personality disorder);
* Anxious and depressive symptoms in the severe range (defined by >27 on the PROMIS Level 2 Anxiety or > 32 on the PROMIS Level 2 Depression);
* Psychological distress symptoms in the severe range (Kessler Psychological Distress Scale [K10] >= 30);
* Threshold scores on pre-screening and follow-up measures exceeded for Mania, Suicidal Ideation, Psychosis, Repetitive Thoughts & Behaviors, Dissociation
* Moderate alcohol, tobacco, or drug use;
* Self-reported diagnosis of neurological condition (e.g., traumatic brain injury, amnesia, epilepsy, stroke, etc.);
* Self-reported presence of any serious medical condition (e.g., cancer, thyroid disorder, multiple sclerosis, etc.);
* Recent bereavement or major loss;
* History of unexplored, untreated traumatic experiences or adverse childhood events.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 860 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Psychological wellbeing | Baseline, Post-intervention (4 weeks), Follow-up (8 weeks)
  Psychological well-being will be assessed using the Warwick-Edinburgh Mental Well-being Scale (WEMWBS), which includes 14 positively worded items of mental well-being for the past 2-weeks, on a 5-point Likert scale from 1 (None of the time) to 5 (All of the time).

SECONDARY OUTCOMES:
Psychological Distress | Baseline, Mid-intervention (2 weeks), Post-intervention (4 weeks), Follow-up (8 weeks)
  Psychological distress will be assessed using the Kessler Psychological Distress Scale (K10), a 10-item self-report measure of psychological distress over the past month, on a 5-point Likert scale from 1 (None of the time) to 5 (All of the time)
Anxiety | Baseline, Mid-intervention (2 weeks), Post-intervention (4 weeks), Follow-up (8 weeks)
  Anxiety will be assessed using (i) the PROMIS Anxiety Short Form, a 7-item measure of the pure domain of anxiety over the past 7 days, on a 5-point Likert scale from 1 (Never) to 5 (Always), and (ii) the Anxiety subscale of the Depression, Anxiety and Stress Scale (DASS-21), a 7-item measure of anxiety over the past 7 days, on a 4-point Likert scale from 0 (Did not apply to me at all - never) to 3 (Applied to me very much, or most of the time).
Depression | Baseline, Mid-intervention (2 weeks), Post-intervention (4 weeks), Follow-up (8 weeks)
  Depression (secondary outcome) will be assessed at T0, T0.5, T1, and T2 using the PROMIS Depression Short Form, an 8-item measure of depression over the past 7 days, on a 5-point Likert scale from 1 (Never) to 5 (Always).
Nonattachment | Baseline, Mid-intervention (2 weeks), Post-intervention (4 weeks), Follow-up (8 weeks)
  Nonattachment will be assessed using the Nonattachment Scale (NAS-7, which measures the Buddhist notion of nonattachment on a 7-point Likert scale from 1 (Disagree strongly) to 5 (Agree strongly).
Trait Mindfulness | Baseline, Mid-intervention (2 weeks), Post-intervention (4 weeks), Follow-up (8 weeks)
  Trait Mindfulness will be assessed with the Five Facet Mindfulness Questionnaire (FFMQ), a 15-item measure that includes five factors representing elements of mindfulness, on a 5-point Likert scale from 1 (Never or very rarely true) to 5 (Very often or always true)
Decentering | Baseline, Mid-intervention (2 weeks), Post-intervention (4 weeks), Follow-up (8 weeks)
  Decentering (secondary outcome) will be assessed at T0, T0.5, T1, and T2 using the Experiences Questionnaire (EQ), an 11-item measure of decentering, on a 5-point Likert scale from 1 (Never) to 5 (All the time).
Equanimity | Baseline, Mid-intervention (2 weeks), Post-intervention (4 weeks), Follow-up (8 weeks)
  Equanimity will be assessed with the Two Factor Equanimity Scale (EQUA-S), a 14-item measure of equanimity, on a 5-point Likert scale from 1 (Never) to 5 (Very often or always).
Repetitive Negative Thoughts | Baseline, Mid-intervention (2 weeks), Post-intervention (4 weeks), Follow-up (8 weeks)
  Repetitive negative thoughts will be assessed with the Repetitive Negative Thoughts Questionnaire (RNTQ), a 22-item measure of repetitive negative thinking, on a 6-point Likert scale from 1 (Not at all typical of me) to 6 (Extremely typical of me)
Emotional Regulation | Baseline, Mid-intervention (2 weeks), Post-intervention (4 weeks), Follow-up (8 weeks)
  Emotional Reactivity will be assessed using the Perth Emotional Reactivity - Short Form (PERS-S), an 18-item measure of the activation, intensity, and duration of one's emotional responses, on a 5-point Likert scale from 1 (Very unlike me) to 5 (Very like me)
Attentional Control | Baseline, Mid-intervention (2 weeks), Post-intervention (4 weeks), Follow-up (8 weeks)
  Attention Control will be assessed with the Attention Control Scale - Short-Form (ATTC-SF), a 10-item measure that includes two subscales of attention (shifting and focusing), on a 4-point Likert scale ranging from 1 (Almost never) to 4 (Always).
Emotional Reactivity | Baseline, Mid-intervention (2 weeks), Post-intervention (4 weeks), Follow-up (8 weeks)
  Emotional Regulation measured by the Perth Emotional Reactivity - Short Form (PERS-S), an 18-item measure of the activation, intensity, and duration of one's emotional responses on a 5-point Likert scale from 1 (Very unlike me) to 5 (Very like me).
Social Anxiety | Baseline, Post-intervention (4 weeks)
  Social Anxiety will be assessed with the Social Anxiety Disorder Severity Scale (SAD-D), a 10-item measure assessing the severity of symptoms of social anxiety in the past 7 days on a 5-point Likert scale from 0 (Never) to 4 (All of the time).
Sleep Quality | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
  Sleep will be measured by the single-item Sleep Quality Scale on a 10-point Likert scale: Terrible (1), Poor (2-4), Fair (5-7), Good (7-9) to Excellent (10)

OTHER OUTCOMES:
Momentary Mood | Daily pre and post meditation session (i.e. Days 1 through 28 excluding 4 rest days)
  Momentary mood will be assessed daily, before and after each meditation session with a modified English version of the Multidimensional Mood Questionnaire (MDMQ). The MDMQ assesses valence, arousal, and calmness dimensions of momentary mood using six items on a 7-point Likert scale (with end-points labelled "very"). Participants will respond to the statement "At this moment I feel:" 1. tired-awake; 2. content-discontent; 3. agitated-calm; 4. energetic-lacking energy; 5. well-unwell; 6. relaxed-tense.
State Mindfulness | 1 of 4 measures randomly assigned on days 1 through 28 excl. rest days (i.e. random assignment occurs on 24 days)
  State mindfulness will be assessed with a brief 6-item version of the State Mindfulness Scale (SMS) on a 5-point Likert scale with options ranging from 1 (Not at all) to 5 (Very well).
Attention | 1 of 4 measures randomly assigned on days 1 through 28 excl. rest days (i.e. random assignment occurs on 24 days)
  Attention will be assessed with the attention regulation and self-regulation subscales of the Multidimensional Assessment of Interoceptive Awareness (MAIA) on a 6-point Likert scale ranging from 1 (Never) to 6 (Always).
Decentering | 1 of 4 measures randomly assigned on days 1 through 28 excl. rest days (i.e. random assignment occurs on 24 days)
  Decentering will be assessed with a brief 5-item version of the Decentering Subscale of the Toronto Mindfulness Scale (TMS) on a 6-point Likert scale ranging from 1 (Not at all) to 6 (Very much).
Mindful Attitudes | 1 of 4 measures randomly assigned on days 1 through 28 excl. rest days (i.e. random assignment occurs on 24 days)
  Mindful attitudes will be assessed using a face-valid selection of: a) TMS items to reflect attitudes of non-judgement (acceptance/allowance) and curiosity; b) a selection of FFMQ non-judgement subscale items to reflect non-judgement (non-evaluative aspect); c) and NAS-7 items to reflect non-attachment using a 5-point Likert scale ranging from 1 (Not at all) to 5 (Very much).

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas T Van Dam, Principal Investigator — University of Melbourne
Locations (1):
- Contemplative Studies Centre, The University of Melbourne, Carlton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant-level de-identified data will be shared via OSF as soon as is reasonably possible.